CLINICAL TRIAL: NCT06220513
Title: Ultrasound-guided Erector Spinae Plane Block Versus Transversus Abdominis Plane Block for Postoperative Analgesia of Adult Patients Undergoing Laparoscopic Appendectomy
Brief Title: Erector Spinae Plane Block Versus TAP Block for Postoperative Analgesia of Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman abdelnaby Mohamed soliman, Assistant lecturer ofAnaesthesia, intensive care and pain management, Ain Shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: laparoscopic appendectomy pain
Record Dates: First submitted 2024-01-06; First posted 2024-01-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-07

CONDITIONS: Laparoscopic Appendectomy
Keywords: transversus abdominis plane block; erector spinae plane block

STUDY DESIGN:
Intervention Model Description: : a double -blinded randomized clinical study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: - Patients will be allocated in two groups using computer-generated table by a person who has access to the computer-generated table but is not involved in data collection or patient management perioperatively. BLock will be given by Anesthesiologist who is not involved in the study.Data collection will be carried out by a person who is completely blinded to the randomization. The person who analyzed the data statistically will not be involved in randomization or data collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (ESP) block group (Active Comparator): the first group (ESP) will be placed in the lateral decubitus position. The ultrasound probe will be placed in longitudinal orientation at the level of the T9spinous process and then moved the probe 3 cm laterally from the midline. The ultrasound landmarks, which included the T9 transverse process and the overlying erector spinae muscle, will be identified. Under complete aseptic conditions, an 80-mm 21-gauge block needle will be inserted in plane at an angle of 30-40° in cranial-to-caudal direction until the tip contacted the T9 transverse process. After hydro-dissection with 3 mL of isotonic saline solution confirmed the correct needle tip position, 20mL of 0.25% bupivacaine will be injected deep to the erector spinae muscle. The same procedure will be repeated with 20mL of 0.25% bupivacaine solution on the contralateral side.
  Interventions: Procedure: erector spinae plane block (ESP)
- Group B TAP block group (Active Comparator): patients who will receive TAP block. A high-frequency ultrasound probe placed transversely, approximately midway between the iliac crest and costal margin shows the three muscle layers of the abdominal wall. A regional block needle can then be inserted anteriorly and slightly away from the probe and carefully advanced until it reaches the transversus plane. In this 'in-plane' technique. The needle and its tip are visualised throughout the procedure, as it enters the transversus plane after piercing the fascial layer below the internal oblique muscle. The needle will be directed toward the transversus abdominis fascia and injected 20 mL of 0.25% bupivacaine between the rectus abdominis and transversus abdominis muscles. The same procedure will be repeated with 20mL of 0.25% bupivacaine solution on the contralateral side.
  Interventions: Procedure: transversus abdominis plane block(TAP)

INTERVENTIONS:
Procedure: erector spinae plane block (ESP) — patients will receive Ultrasound-guided erector spinae plane block (ESP) block for postoperative analgesia of adult patients undergoing laparoscopic appendectomy.
  Arms: Group A (ESP) block group
Procedure: transversus abdominis plane block(TAP) — patients will receive Ultrasound-guided transversus abdominis plane block(TAP) Block for postoperative analgesia of adult patients undergoing laparoscopic appendectomy.
  Arms: Group B TAP block group

SUMMARY:
Laparoscopic appendectomy is the most frequently performed surgery in patients who develop acute appendicitis. This surgical technique is more advantageous than an open appendectomy in terms of fewer complications, less postoperative pain, and a faster return to normal daily activities. Even though the laparoscopic technique is minimally invasive, postoperative pain is inevitable. Furthermore, it may affect the patients' mobility and cause them to stay in the hospital for a more extended period .The study aimed to compare the effectiveness and the safety of ultrasound-guided erector spinae plane block versus ultrasound-guided transversus abdominis plane block (TAP) as postoperative analgesia methods after laparoscopic appendectomy.

DETAILED DESCRIPTION:
Acute appendicitis develops in a progressive and irreversible manner, even if the clinical course of acute appendicitis can be temporarily modified by intentional medications. Reliable and real-time diagnosis of acute appendicitis can be made based on findings of the white blood cell count and enhanced computed tomography. Emergent laparoscopic appendectomy is considered as the first therapeutic choice for Acute appendicitis .

The reported advantages of laparoscopic appendectomy compared with open appendectomy are less postoperative pain, less wound infection, and better cosmetic results. Even though the laparoscopic technique is minimally invasive, postoperative pain is inevitable. Furthermore, it may affect the patients' mobility and cause them to stay in the hospital for a more extended period .An intraperitoneal injection of local anesthetics is one of the analgesic modalities that are used to control pain in such cases but it is insufficient analgesic in most of patients and has short duration effect .

Recently Ultrasound-guided nerve blocks were effectively used for postoperative analgesia in different types of surgical procedures .Both erector spinae plane block and oblique subcostal transversus abdominis plane block have been used effectively to reduce pain after laparoscopic appendectomy.

In ultrasound-guided Transversus Abdominis Plane (TAP) Block local anesthetic (LA) is deposited in the plane between the transversus abdominis and posterior sheath of the rectus muscle in approximately midway between the iliac crest and costal margin .To anesthetize The terminal branches of the lower six thoracic and first lumbar nerve lie within, providing analgesia of the anterior and lateral abdominal wall .This block has a low risk for serious complications such as bowel or diaphragm perforation and lacerations of the liver. Abdominal wall hematoma, vascular injury, and local anesthetic toxicity are also potential but rare complications . Owing to safety of ultrasound-guided needle placement a 'real-time' visualization through dynamic scanning is used .

The ultrasound-guided Erector Spinae Plane (ESP) block is a paraspinal fascial plane block in which local anesthetic is administered between the erector spinae muscle and the thoracic transverse processes at the levels of the T7-T9 transverse processes, resulting in spread between the T6 and T12 segmental levels, blocking the dorsal and ventral rami of the abdominal spinal nerves.

This blockage of the dorsal and ventral rami of the spinal nerves helps to achieve a multi-dermatomal sensory block of the anterior, posterior, and lateral abdominal walls.

ESP block Complications such as vascular puncture, pleural puncture and pneumothorax are the primary complications .Also local anethetic toxicity, infection at needle insertion site and allergy also can occur .

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic appendectomy,
* Patients aged 18-50 years,
* American Society of Anaesthesiologists (ASA) physical status I or II.

Exclusion Criteria:

* Declined informed consent.
* Allergy to local anesthetics.
* Conversion of the laparoscopic surgery to open appendectomy.
* Coagulation disorder.
* Pregnancy,
* BMI more than 40 kg/m2,
* Respiratory disease, liver or kidney disease; and heart disease (heart block, Rheumatic heart or myocardial ischemia).
* Psychiatric problems, that results in lack of communication ability.
* Chronic alcoholism, drug abuse,
* Infection in the area where the block will be applied.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
a numerical rating scale (NRS) | Patients will be asked to record their level of pain at 30 minutes as well as at two, four, six, eight, 12, 18 and 24 hours postoperatively.
  an 11-point scale where 0 indicates no pain and 10 indicates the worst imaginable pain. Patients will chose a whole number to express the degree of their pain both at rest and when moving.

SECONDARY OUTCOMES:
Intraoperative heart rate | the duration of surgery
  Heart rate (HR)in beat per minute will be recorded every 5 min till the end of the surgery.
Incidence of complications | the duration of surgery
  Including nerve injury, hematoma formation, Local anesthetic toxicity, and intravascular injections;
the cumulative consumption of pethidine | the first 24 postoperatively
  At a NRS pain scores of five or above, 50 mg of intravenous pethidine was administered. The total dose of analgesics administered during the first 24 hours will be carefully recorded.
The duration of time before the first request for rescue analgesia post-surgically. | first postoperative hour
  The maximum allowed dose of pethidine will be set at 5 mg/kg/24 h based on lean body weight. The blocks will be considered as failed blocks if patients require more than two doses of rescue analgesia in the first postoperative hour.
intraoperative blood pressure monitoring | the duration of surgery
  mean arterial pressure (MAP) in millimeter mercury will be recorded every 5 min till the end of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Fathy, MD, Study Director — Ainshams university; Mohsen Basyoni, MD, Study Chair — Ainshams university
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Kuscu Y, Gumus Demirbilek S. Ultrasound-guided erector spinae plane block versus oblique subcostal transversus abdominis plane block for postoperative analgesia of adult patients undergoing laparoscopic cholecystectomy: Randomized, controlled trial. J Clin Anesth. 2019 Nov;57:31-36. doi: 10.1016/j.jclinane.2019.03.012. Epub 2019 Mar 6. PMID 30851501
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Sertcakacilar G, Yildiz GO. Analgesic efficacy of ultrasound-guided transversus abdominis plane block and lateral approach quadratus lumborum block after laparoscopic appendectomy: A randomized controlled trial. Ann Med Surg (Lond). 2022 Jun 14;79:104002. doi: 10.1016/j.amsu.2022.104002. eCollection 2022 Jul. PMID 35860161
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Background] Yu N, Long X, Lujan-Hernandez JR, Succar J, Xin X, Wang X. Transversus abdominis-plane block versus local anesthetic wound infiltration in lower abdominal surgery: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2014 Dec 15;14:121. doi: 10.1186/1471-2253-14-121. eCollection 2014. PMID 25580086